CLINICAL TRIAL: NCT04383886
Title: Evaluation of Emergency Department (ED) Staff Stress Level During COVID-19 Pandemic
Acronym: COVER-PRO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0330
Record Dates: First submitted 2020-05-08; First posted 2020-05-12 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Emergency Department Staff During the COVID-19 Pandemic; Emergency Department Staff's Level of Stress
Keywords: COVID-19 pandemic; level of stress; emergency department staff
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emergency department staff
  Interventions: Other: stress and anxiety questionnaire

INTERVENTIONS:
Other: stress and anxiety questionnaire — Emergency department staff will be asked to fill in questionnaires in order to measure their stress and anxiety level, their propensity to have a burn-out, their consumption of psychoactive substances such as alcohol, tobacco, coffee or anxiolytic, their sleep disorder.

SUMMARY:
In the context of the COVID-19 pandemic, Emergency Department (ED) are in front line for the reception of patients presenting COVID-19 symptoms and have to face a new situation given the expected number of patients. Staff participate in suspect patients triage, in the diagnosis and the management of Covid-19 patients, having to follow the instructions and recommendations that evolve in real time, depending on the stage, resources and means available. This situation requires that the staff immediately adaptation within this reorganization and redeployment of the activity. Then; they are subject to many stress and anxiety factors such as:

* Increased activity: massive influx of patients, overload of work, lack of material and human resources
* Modification of practices: training in procedures, measures isolation and prevention of contamination of other patients, replacement by professionals reassigned from other departments
* Ethical dilemma: decisions to be made in an emergency, patient prioritization
* Numerous, evolving information, from various sources and sometimes contradictory (national, governance, service, media)
* Individual: fear of personal contamination and of those close to you, personal organization in a situation of confinement of the population, loss of usual social support
* Anxiety and stress management of patients and relatives, their entourage and colleagues In this study, it is proposed to study the psychic impact of the COVID-19 pandemic on emergency department staff.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* medical and paramedical staff working the the emergency room permanently or specifically during the COVID19 pandemic
* not opposed to participate to this study

Exclusion Criteria:

* Staff under legal protection
* refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency department staff
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-09-12 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Change of emergency department staff's level of stress during the covid19 pandemic, measured using the Chamoux et Simard visual analogic scale | Every 15 days from baseline to 3 months
  The level of stress will be measured using the Chamoux et Simard visual analogic scale. This scale is composed of 3 subscales evaluating the stress level at work, at home and in the life in general. Each scale are rating from 0 to 10, 0 being the absence of stress and 10 the highest level of stress ever experienced a cotation at each scale greater than 6 will defined the presence of a stress.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - SAMU Hospices Civils de Lyon, Lyon
  - Service d'accueil des urgences, Hôpital Edouard Herriot, Hospices Civlis de Lyon, Lyon
  - Service d'accueil des urgences, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Service d'accueil des urgences, Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Hôpital de Villefranche-sur-Saône, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Douplat M, Subtil F, Termoz A, Jacquin L, Verbois F, Potinet V, Hernu R, Landel V, Mazza S, Berthiller J, Haesebaert J, Tazarourte K. Mental Health Consequences of the COVID-19 Outbreak Among Emergency Department Healthcare Workers. Biomed Res Int. 2024 Sep 9;2024:8871959. doi: 10.1155/2024/8871959. eCollection 2024. PMID 39286281
- [Derived] Douplat M, Termoz A, Subtil F, Haesebaert J, Jacquin L, Durand G, Potinet V, Hernu R, Nohales L, Mazza S, Berthiller J, Tazarourte K. Changes over time in anxiety, depression, and stress symptoms among healthcare workers in French emergency departments during the first COVID-19 outbreak. J Affect Disord. 2022 Nov 1;316:194-200. doi: 10.1016/j.jad.2022.08.028. Epub 2022 Aug 15. PMID 35981626